CLINICAL TRIAL: NCT04827030
Title: A Double-blind Randomized Non-inferiority Trial of Erector Spinae Block (ESP) Versus Paravertebral Block (PVB) Before Breast Cancer Surgery: Effects on Acute Postoperative Pain.
Brief Title: ER-One: A Double-blind Trial of Erector Spinae Block (ESP) Versus Paravertebral Block (PVB) Before Breast Cancer Surgery
Acronym: ER-One
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IC 2020-04
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Surgery
Keywords: Breast; Surgery; anaesthetics
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: A Double-blind Randomized non-inferiority Trial of erector spinae block (ESP) versus paravertebral block (PVB)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine hydrochloride injected by Erector Spinae block (Active Comparator): The injection will be performed with Ropivacaine hydrochloride 0.6 ml/kg of solution at 5 mg/ml up to 30 ml
  Interventions: Drug: Ropivacaïne Hydrochloride by Erector Spinae block
- Ropivacaine hydrochloride injected by Paravertebral block (Active Comparator): The injection will be performed with Ropivacaine hydrochloride 0.6 ml/kg of solution at 5 mg/ml up to 30 ml
  Interventions: Drug: Ropivacaïne Hydrochloride by Paravertebral block

INTERVENTIONS:
Drug: Ropivacaïne Hydrochloride by Erector Spinae block — Ropivacaïne Hydrochloride Erector Spinae puncture will be performed with ultrasound guidance. Then 0.50% Ropivacaine hydrochloride will be injected at a dose of 0.6 ml/kg of actual weight, without exceeding 30 ml.
  Other Names: Naropin
  Arms: Ropivacaine hydrochloride injected by Erector Spinae block
Drug: Ropivacaïne Hydrochloride by Paravertebral block — Paravertebral puncture will be performed with ultrasound guidance. Then 0.50% Ropivacaine hydrochloride will be injected at a dose of 0.6 ml/kg of actual weight, without exceeding 30 ml.
  Other Names: Naropin
  Arms: Ropivacaine hydrochloride injected by Paravertebral block

SUMMARY:
The block (ESP or PVB) will be performed preoperatively in the recovery room under standard monitoring. After setting a peripheral venous access, patient will be installed on lateral decubitus position on the opposite side of the block.

DETAILED DESCRIPTION:
The block will be performed with IV Remifentanil sedation Target-Controlled Infusion mode at 2ng/ml and oxygen therapy.

For the erector spinae plane block:

The puncture will be performed with ultrasound guidance. The ultrasound probe will be placed parallel to the spine parasagittally at the T3 transverse process level. The needle will be introduced and visualized to the plane of the ultrasound image ("in plane").

The desired injection site is between the fascia of the erector muscle of the spine and the transverse process at the T3 level. The operator ensures the correct localization of the needle with saline solution. Then 0.50% Ropivacaine hydrochloride will be injected at a dose of 0.6 ml/kg of actual weight, without exceeding 30 ml.

For paravertebral block:

The T2 intervertebral space will be located by identifying compared to C7, a prominent cervical vertebra, or by ultrasound by counting the thoracic vertebrae from the first rib. The paravertebral space will be identified by placing the ultrasound probe in a parasagittal or transverse position. The needle will go through the paravertebral muscles and the costo-transverse ligament or by a latero-medial approach using ultrasound. The block will be performed using a 22-gauge 8cm long needle. When the paravertebral space has been reach, an aspiration test will be performed and then 0.6 ml/kg of solution (Ropivacaine hydrochloride solution at 5 mg/ml up to 30 ml) will be injected.

ELIGIBILITY:
Inclusion Criteria:

1. Woman with breast adenocarcinoma without metastasis or breast in situ adenocarcinoma (with or without breast reconstruction by prosthesis) to by treated:

   * either by breast-conserving surgery with axillary dissection,
   * either by modified radical mastectomy with axillary dissection
   * either by modified radical mastectomy with lymph node dissection
   * either by modified radical mastectomy without axillary
2. Patients aged between 18 and 85 years old.
3. ASA class 1, 2 or 3 (Physical Status Classification System of American Society of Anesthesiologists (ASA)).
4. Signed informed consent form.
5. Patient able to answer self-assessment questionnaires (sufficient understanding of evaluations and in French).
6. Patient affiliated to the health care insurance.

Exclusion Criteria:

1. Preoperative consumption of opioid in the patient's current medications within three months before inclusion.
2. Ipsilateral breast surgery during 3 months prior to the inclusion.
3. Allergy to local anaesthetics and morphine and NSAID.
4. Local skin inflammation at the puncture area.
5. Bilateral breast surgery planned at inclusion.
6. Major immediate ipsilateral breast reconstruction by using tissue flap procedure (example: latissimus dorsi flap, Deep Inferior Epigastric Perforator (DIEP), Transverse Rectus Abdominis Musculocutaneous (TRAM)…).
7. Any contra-indication or patient's refusal for regional anesthesia.
8. Male subjects.
9. Pregnant woman or breastfeeding.
10. B blocker medication.
11. Patient already participating in an analgesia protocol that may interfere with the pain assessment criteria.
12. Patient under legal protection.
13. Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Comparison of ESP versus PVB on acute postoperative pain | 24 hours
  Percentage of patients needed morphine during the first two postoperative hours in each treatment arm

SECONDARY OUTCOMES:
Postoperative morphine consumption | 2 hours
  Dose of opioid, in the Post-Anesthesia Care Unit (PACU)
Consumption of remifentanil in the Operating Room (OR) | During the period from the surgical incision to the end of the surgical dissection
  Dose of Remifentanil during the Operating Room (OR) period
Acute early postoperative pain by Visual Analog Scale (VAS) | 24 hours
  VAS (no pain=0, worst pain=10) at arrival in the PACU, every 30 minutes in the Post-Anaesthesia Care Unit (PACU), VAS at 4 and 24 hours. Pain scores will be evaluated at rest and after shoulder movement
Percentage of nausea or vomiting | 2 hours
  Number of patient who related nausea or vomiting side effects will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 5.0)
Incidence of complications and side effects of each block | 30 days
  Complications and side effects of each block will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 5.0)
Post-operative extend of dermatomes blocked | 2 hours
  The extent of dermatomes blocked as measured by clinical examination to determine area where temperature perception change

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FUMOLEAU, PhD, Study Director — Institut Curie; Julien RAFT, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (5):
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - AP-HP Hôpital Tenon, Paris
  - Institut Curie, Saint-Cloud
  - Institut Claudius Régaud UICT, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Raft J, Dureau S, Fuzier R, Auge M, Lamotte AS, Lemoine A, Albi-Feldzer A. Erector spinae plane block versus paravertebral block for major oncological breast surgery: a multicentre randomised controlled trial. Br J Anaesth. 2025 Sep;135(3):772-778. doi: 10.1016/j.bja.2025.05.051. Epub 2025 Jul 24. PMID 40707285